CLINICAL TRIAL: NCT05355883
Title: Effects of Remote Ischemic Conditioning on Bimanual Skill Learning, Bimanual Coordination, and Corticospinal Excitability in Children With Unilateral Cerebral Palsy
Brief Title: Remote Ischemic Conditioning, Bimanual Skill Learning, and Corticospinal Excitability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Swati Manoharrao Surkar, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-001913
Record Dates: First submitted 2022-01-15; First posted 2022-05-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Unilateral Cerebral Palsy; Hemiplegic Cerebral Palsy; Remote Ischemic Conditioning
Keywords: Cerebral palsy; Bimanual coordination; Corticospinal excitability
MeSH Terms: conditions — Cerebral Palsy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are masked to group assignment (RLIC vs. Sham conditioning) and the assessor will be masked to group assignment of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (RIC) (Experimental): RIC is achieved via blood pressure cuff inflation to at least 20 mmHg above systolic blood pressure to 250 mmHg on the more involved arm. RIC involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. RIC is performed on visits 2-6.
  Intervention
  * Hand Arm Bimanual Intensive Therapy (HABIT)
  * Bimanual cup stacking training
  * Balance training
  Interventions: Behavioral: Remote Ischemic Conditioning (RIC); Behavioral: Hand Arm Bimanual Intensive Therapy (HABIT); Behavioral: Bimanual Cup Stacking Training; Behavioral: Balance training
- Sham Conditioning (Sham Comparator): Sham conditioning is achieved via blood pressure cuff inflation to 25 mmHg on the more involved arm. RIC involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. RIC is performed on visits 2-6.
  Intervention
  * Hand Arm Bimanual Intensive Therapy (HABIT)
  * Bimanual cup stacking training
  * Balance training
  Interventions: Behavioral: Sham conditioning; Behavioral: Hand Arm Bimanual Intensive Therapy (HABIT); Behavioral: Bimanual Cup Stacking Training; Behavioral: Balance training

INTERVENTIONS:
Behavioral: Remote Ischemic Conditioning (RIC) — See descriptions under arm/group descriptions. RIC is delivered for 5 intervention visits. Visits 1 is the pre-training assessment visit, visits 2-6 are RIC plus training visits, visit 7 is a post-training assessment visit.
  Other Names: Remote limb ischemic conditioning
  Arms: Remote Ischemic Conditioning (RIC)
Behavioral: Sham conditioning — See descriptions under arm/group descriptions. Sham conditioning is delivered for 5 intervention visits. Visits 1 is the pre-training assessment visit, visits 2-6 are RIC plus training visits, visit 7 is a post-training assessment visit.
  Other Names: Sham
  Arms: Sham Conditioning
Behavioral: Hand Arm Bimanual Intensive Therapy (HABIT) — HABIT is a child-friendly, intensive intervention directed at improving bimanual coordination and function of the affected arm. The intervention employed in this study includes various age-appropriate fine and gross motor bimanual activities that will be delivered in a play context. Children practice bimanual activities for 6 hours per day, 5 days per week, for 1 week.
  Other Names: Bimanual skill training
Behavioral: Bimanual Cup Stacking Training — Children practices bimanual cup stacking, 15 trials/day for 5 consecutive day.
  Other Names: Cup stacking task
Behavioral: Balance training — All children undergo training on a balance board, learning to hold the board level with equal weight on each leg and using various bilateral upper extremity strategies. Participants perform the balance task for 15, 30-second trials per day at visits 2-6.

SUMMARY:
Unilateral cerebral palsy (UCP) is a leading cause of childhood disability. An early brain injury impairs the upper extremity function, bimanual coordination, and impacts the child's independence. The existing therapeutic interventions have higher training doses and modest effect sizes. Thus, there is a critical need to find an effective priming agent to enhance bimanual skill learning in children with UCP. This study aims to determine the effects of a novel priming agent, remote ischemic conditioning (RIC), when paired with intensive bimanual skill training to enhance bimanual skill learning and to augment skill dependent plasticity in children with UCP.

DETAILED DESCRIPTION:
Ischemic conditioning (IC) is a phenomenon of protecting the target organ from ischemia by directly exposing it to brief episodes of sublethal ischemia. RIC is a clinically feasible way of performing IC where episodes of ischemia and reperfusion are delivered with cyclic inflation and deflation of a blood pressure cuff on the arm or leg. Pre-clinical and preliminary clinical trials in humans show neuroprotective effects of RIC. Investigators prior work has shown that when paired with motor training, RIC enhances motor learning in healthy individuals. Based on these diversified benefits of RIC, the central hypothesis is that the multifactorial mechanisms of RIC can be harnessed as a priming agent to enhance motor learning and augment neuroplasticity in children with UCP. The Specific Aims are: 1) to determine the effects of RIC + training on bimanual skill performance, and 2) to determine the effects of RIC + training on corticospinal excitability in children with UCP. In this triple blind, randomized controlled trial, 30 children with UCP, ages 6-16 years will first undergo bimanual speed stack performance, functional upper extremity, and Transcranial Magnetic Stimulation assessments. Children will then undergo RIC/Sham conditioning plus training. Investigators will deliver RIC/sham conditioning via cyclic inflation and deflation of a pressure cuff on the paretic arm using a standard protocol. Training will involve 5 days (15 trials/day) of bimanual speed stack training and intensive bimanual training using hand arm bimanual intensive therapy (HABIT) with a standard dose of 6 hours/day for 5 days. The children will perform the same baseline assessments post-intervention. Investigators hypothesize that compared to sham conditioning + training, RIC + training will significantly enhance: 1) bimanual skill performance (decrease in movement time (sec) to complete bimanual speed stack task), 2) bimanual function (increase in the Assisting Hand Assessment scores), 3) cortical excitability in the ipsilesional primary motor cortex (M1) (larger amplitude of motor evoked potentials and lower resting or active motor thresholds), and 4) reduce motor cortex inhibition (reduced short-interval intracortical inhibition and increase in intracortical facilitation in ipsilesional M1). The long-term goal is to develop effective interventions to improve function of children with UCP. Outcomes of this project will provide critical ingredients for designing Phase II trials that will determine the effects of RIC combined with different dose of intensive behavioral interventions to improve functional outcomes in children with UCP.

ELIGIBILITY:
Inclusion Criteria:

Children diagnosed with unilateral cerebral palsy, ages 6-16 years

* Manual Ability Classification System (MACS) levels I-III
* Ability to complete a stack of 3 cups in 2 minutes
* Mainstream in school and has sufficient cognition to follow the experiment instructions

Exclusion Criteria:

* Children with other developmental disabilities such as autism, developmental coordination disorders, etc.

  * Children with absent active motor threshold
  * Children with cognitive deficits or communication problem
  * Children with known cardiorespiratory and vascular dysfunctions
  * Children with metabolic disorders, neoplasm, hydrocephalus
  * Children who are receiving other adjunct therapies such as rTMS and tDCS
  * Children with seizures and on anti-seizure medications
  * Children with metal implants and incompatible medical devices for MRI scans

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Assisting Hand Assessment | Baseline and 1 week
  Assisting Hand Assessment assesses bimanual coordination and affected hand function. A 5-point change from pre- to post-intervention is considered a clinically meaningful improvement.
Change in Bimanual Task Performance | Baseline and 1 week
  The time (seconds) to complete each trial of cup stack, which will be averaged across three trials. This will be measured at visit 1 (pre-) and visit 7 (post-intervention). Smaller time to complete the task indicates better performance.
Change in Resting and Active Motor Thresholds | Baseline and 1 week
  The minimum intensity of the stimulator output required to produce an MEP of > 50 μV will be determined using maximum-likelihood parameter estimation by a sequential testing (ML-PEST) algorithm from the lesioned and non-lesioned cortex. Greater reduction in resting and active motor threshold from pre- to post-intervention indicates greater corticospinal excitability.
Change in Stimulus-response curves | Baseline and 1 week
  Suprathreshold intensities of 110%, 120%, 130%, 140%, and 150% of resting motor threshold will be administered randomly on the lesioned and non-lesioned cortex. Greater motor evoked potential response at each of these intensities indicate greater corticospinal excitability.

SECONDARY OUTCOMES:
Change in Box and Blocks Test (BBT) | Baseline and 1 week
  BBT is a standard test to assess manual speed. Greater number of blocks transferred indicates greater manual speed.
Change in Nine Hole Peg Test (NHPT) | Baseline and 1 week
  NHPT is a standard test to assess manual speed and dexterity. Smaller time to complete NHPT indicates greater speed and dexterity.
Change in Jebsen Hand Function Test (JHFT) | Baseline and 1 week
  JHFT assesses fine and gross hand and arm movements. Smaller time to complete JHFT indicates better hand function.
Change in Balance performance | Baseline and 1 week
  The average amount of time in seconds that a participant maintains the stability platform within ±5° of horizontal position during 15 trials of 30 seconds each. The total score will range between 0-30 seconds. Higher balance score indicates better balance performance. Greater average balance time indicates better balance performance.
Change in Hand grip and pinch strength | Baseline and 1 week
  Hand grip and pinch strength assesses hand muscle strength. Greater hand and pinch strength indicates greater strength of hand muscles.
Change in Short-Interval Intracortical Inhibition (SICI) | Baseline and 1 week
  For SICI, a subthreshold (80% RMT) conditioning pulse to the motor hotspot will be applied followed by a suprathreshold (120% RMT) test pulse 3 milliseconds later. Reduction in SICI indicates intracortical facilitation.
Change in Intracortical Facilitation (ICF) | Baseline and 1 week
  For ICF, the interstimulus interval will increase to 12 milliseconds. Greater ICF indicates greater intracortical facilitation.
Change in accelerometry derived variables | Baseline and 1 week
  Number of movements, use ratio, magnitude ratio, bilateral magnitude, and acceleration variability will be quantified using wrist worn accelerometers. Greater values indicate better bimanual performance.

CONTACTS AND LOCATIONS:
Overall Officials: Swati Surkar, Principal Investigator — East Carolina University
Locations (1):
- Dept. of Physical Therapy, East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on NIH figshare network and will be made available on request.
Supporting Information: ICF
Time Frame: After publishing the results of the study
Access Criteria: Data will be made available upon request to the principal investigator.

REFERENCES:
- [Background] Surkar SM, Hoffman RM, Willett S, Flegle J, Harbourne R, Kurz MJ. Hand-Arm Bimanual Intensive Therapy Improves Prefrontal Cortex Activation in Children With Hemiplegic Cerebral Palsy. Pediatr Phys Ther. 2018 Apr;30(2):93-100. doi: 10.1097/PEP.0000000000000486. PMID 29578992
- [Background] Dirnagl U, Becker K, Meisel A. Preconditioning and tolerance against cerebral ischaemia: from experimental strategies to clinical use. Lancet Neurol. 2009 Apr;8(4):398-412. doi: 10.1016/S1474-4422(09)70054-7. PMID 19296922
- [Background] Gidday JM. Cerebral preconditioning and ischaemic tolerance. Nat Rev Neurosci. 2006 Jun;7(6):437-48. doi: 10.1038/nrn1927. PMID 16715053
- [Background] Stetler RA, Leak RK, Gan Y, Li P, Zhang F, Hu X, Jing Z, Chen J, Zigmond MJ, Gao Y. Preconditioning provides neuroprotection in models of CNS disease: paradigms and clinical significance. Prog Neurobiol. 2014 Mar;114:58-83. doi: 10.1016/j.pneurobio.2013.11.005. Epub 2014 Jan 2. PMID 24389580
- [Background] Kharbanda RK, Nielsen TT, Redington AN. Translation of remote ischaemic preconditioning into clinical practice. Lancet. 2009 Oct 31;374(9700):1557-65. doi: 10.1016/S0140-6736(09)61421-5. PMID 19880021
- Available data/document: Informed Consent Form — https://epirate.ecu.edu/App/app/portal/smartform/read?project=com.webridge.entity.Entity%5BOID%5B21688D0E003911ECFE80AAA590565000%5D%5D&projectEditorView=com.webridge.entity.Entity%5BOID%5BDB15548F56BE6942A0B8A537449C64C3%5D%5D